CLINICAL TRIAL: NCT06294002
Title: Effect of Different Neuromuscular Training Modalities on Postural Stability in Healthy Recreation People: A Randomised Controlled Trial
Brief Title: Neuromuscular Training & Postural Stability
Acronym: STABLEFIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Novi Sad (Other)
Responsible Party: Principal Investigator, Dragan Marinkovic, Lead Investigator, University of Novi Sad
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 46-06-04/2020-1
Record Dates: First submitted 2024-02-20; First posted 2024-03-05 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Postural Stability
Keywords: postural control; exercise; vibration training; balance; neuromuscular adaptation
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Dynamic neuromuscular stabilization group (DNS) (Experimental): DNS - Dynamic neuromuscular stabilization intervention
  Interventions: Other: Dynamic neuromuscular stabilisation group
- Whole body vibration group (VIBRO) (Experimental): VIBRO - Whole body vibration intervention
  Interventions: Other: Whole body vibration group
- Dynamic neuromuscular stabilisation with whole body vibration group (MIX) (Experimental): MIX group - neuromuscular and whole body vibration intervention
  Interventions: Other: Dynamic neuromuscular stabilisation with whole body vibration group
- Control group (CONTROL) (No Intervention): Control group - no intervention

INTERVENTIONS:
Other: Dynamic neuromuscular stabilisation group — DNS group protocol involved 5 min a moderate intensity warm-up, 40 minutes of DNS movements according to the DNS approach, different diaphragmatic breathing, mobility and controlled movement exercises and 5 minutes of cool-down. Exercises gradually increased in complexity and difﬁculty level regarding DNS training principles. The participants were instructed to refrain from engaging in high-intensity anaerobic or anaerobic resistance training throughout the study period to prevent potential disruptions in the study results.
  Arms: Dynamic neuromuscular stabilization group (DNS)
Other: Whole body vibration group — WBV was performed on the Power Plate Next Generation vibration platform (Power Plate North America, Chicago, IL). All training routines were approximately 50 minutes long, commencing with 5 minutes of moderate-intensity warm-up and concluding with a cool-down period. The program consisted of 8-10 static and dynamic exercises for PS that progressively increased in difficulty and complexity. During the training process, the frequency increased from 20 to 35 Hz in the last week of the experiment; the exercise duration was from 20 - 60 seconds (in the previous week), followed by 1-minute seated rest. Moreover, the complexity and difficulty of exercise increased over the experimental period. The resting period between sets was constant from the start to the end of the training process. During the experiment, the WBV intervention group performed three weekly training sessions.
  Arms: Whole body vibration group (VIBRO)
Other: Dynamic neuromuscular stabilisation with whole body vibration group — The MIX group underwent a two-month training program consisting of three weekly sessions, including a 50-minute exercise program with a 5-minute warm-up and cool-down period. The training included 20 minutes of WBV and 20 minutes of DNS training, following previous research and training recommendations. VIBRO exercises were performed on the Power Plate Next Generation vibration platform, with 6-8 exercises for balance and PS. Participants were advised not to engage in high-intensity anaerobic or anaerobic resistance training. The training protocol was adapted from previous research.
  Arms: Dynamic neuromuscular stabilisation with whole body vibration group (MIX)

SUMMARY:
Background: Postural stability (PS) is a vital function that helps maintain equilibrium during standing still, locomotion, and any activities requiring high balance performance. Under static and dynamic conditions, PS is a fundamental factor for the quality of movement in everyday activities or sports. PS and adaptive ability are required in sports due to the interactions between the sensory and motor systems, which regulate postural adjustments by processing information from the visual, vestibular, and somatosensory systems, as reported by previous studies. The interest in using different exercises and protocols for improving PS in sports and physiotherapy has grown in the last few decades. Experts have proposed various training modalities to increase neuromuscular stability, balance, postural control, and general stability. Dynamic Neuromuscular Stabilization (DNS) is a complex of correction exercises with a neuromuscular approach based on improving breathing, fundamental movements, and principles of developmental kinesiology. Whole body vibration training (WBV) is a neuromuscular training approach that has recently become very popular among researchers and practitioners in health and sport. It is usually used as an additional method in a conventional training routine. Designing the training program to achieve the optimal benefits for PS in healthy young adults is important in general personal health management. Although different training protocols have improved PS and general stability in everyday activities, there is still considerable debate regarding the optimal exercise modalities within an exercise program. Aim: The purpose of this study is to determine the effects of dynamic neuromuscular stabilisation (DNS), whole-body vibration (WBV), and a combination of DNS and WBV (MIX) training modalities on postural stability (PS) in healthy recreation participants. Method and materials: 180 gender-balanced groups were divided into four groups, MIX, DNS, VIBRO and CONTROL and underwent two months of treatment. The single and double-leg Center of Force (COF) parameters were collected on the Forceplate.

DETAILED DESCRIPTION:
Study design The purpose of this study is to determine the effects of dynamic neuromuscular stabilisation (DNS), whole-body vibration (WBV), and a combination of DNS and WBV (MIX) training modalities on postural stability (PS) in healthy recreation participants. The study presents an Interventional study to improve postural stability, and the main objective is prevention. The study model is parallel with four groups.

Participants The randomised, controlled interventional trial enrolled a gender-balanced group of 180 healthy young participants. The initial sample of respondents was recruited through an open online application that lasted two months (from 10.2.2022. to 10.4.2022.) (n=250), after which the first selection of respondents was started (n=230). Recruitment was completed after the optimal sample of subjects was filled (15.4.2022). The study sample was divided using stratified randomisation into the MIX group (n = 58), DNS group (n=57), VIBRO (n=57), and CONTROL group (n=58). At the end of the experimental program, the final sample was 180 (MIX=45; DNS=45; VIBRO=44; CONTROL=43). When stratifying, researchers use proportionate sampling to maintain the correct proportions of genders in every group. After explaining the experimental protocol, each subject provided written informed consent before participating in the study, per the Declaration of Helsinki and the Novi Sad University Human Research Ethics Committee guidelines (ethical approval number: 46-06-04/2020-1). The interventional program was conducted from 25.4.2022. to 25.6.2022. Ethics committee - commission for the implementation of scientific project research.

The exclusion criteria were:

* history of neurological or musculoskeletal disorders;
* clinical conditions that could impair balance (motor disorders, medical conditions like diabetes, heart disease, stroke, issues with vision, thyroid, nerves, or blood vessels).

The inclusion criteria for this study were:

• the absence of injuries in the past six months and the absence of other medical conditions, including COVID-19, no programmed physical activity in the past three months.

Testing procedures The testing was conducted at the Faculty of Sport and Physical Education, University of Novi Sad, Serbia. All participants were tested in the morning before their training session in indoor environmental conditions (temperature: 18-21°C; relative humidity: 40-60%). Before starting a performance task, general information about the examinees was recorded, including gender, age, height, and mass. Participants were instructed to wear minimal clothing and remove all footwear for height and mass measurements. In addition, they were required to eat and drink sparingly and void their bladder/excrete as needed before presenting for assessment. A stadiometer (0.1 cm accuracy, SECA Instruments Ltd, Hamburg, Germany) is a secondary outcome for height and mass measurements. Initial testing was conducted on 20.4.2022 and final on 25.6.2022.

Static PS was assessed with a laboratory-grade 0.5 m Footscan® plate (RSscan International, Lammerdries, Belgium) with 4096 sensors and a scanning rate of up to 300 Hz. The subject performed an individual single and double-leg task with three trials, each lasting 30 seconds with a two-minute break between each trial. During the double-leg stance test, participants were instructed to maintain an upright posture as still as possible. They were asked to stand in their natural, comfortable position with their eyes open and fixed on a cross positioned at approximately eye level on a blackboard 5 meters away. Participants stood barefoot with their feet placed shoulder-width apart on a platform, and their arms were kept by their sides. Each participant was required to maintain this stable posture, and measurement started after 10 seconds (preparation period to avoid transient effects). During the single-limb stance test, participants were instructed to balance on one foot. This foot was positioned to point directly forward, aligning with reference lines in the frontal and sagittal planes. The swinging leg was flexed at the hip and knee joints to approximately 90 degrees while both arms hung naturally and relaxed at their sides. Participants were further instructed to maintain as steady a posture as possible, focusing their gaze straight ahead on a point situated 65 centimetres away on the wall. The order of testing between the left and right legs was randomised. Each participant was required to maintain this stable position, and measurement started after 5 seconds (preparation period to avoid transient effects).

Tests for static PS were the gold standard in measuring balance and were used to obtain biomechanical parameters of static PS. All measurements were performed in triplicate, and the mean score was retained for subsequent evaluations and analyses. The sequence of performing the balance tasks was randomised.

The software calculated the single and double-leg Sway Area (cm²), Center of Force (COF) travelled way (mm), Medio-Lateral (ML) displacement (mm), and Anterior-Posterior (AP) displacement (mm) as primary outcomes. As stated in previous research, the following protocol was chosen based on their varying difficulty and everyday use and is cited as reliable.

Interventions Dynamic neuromuscular stabilisation group (DNS) The DNS group's protocol involved 5 min a moderate-intensity warm-up, 40 minutes of DNS movements according to the DNS approach, different diaphragmatic breathing, mobility and controlled movement exercises and 5 minutes of cool-down. Exercises gradually increased in complexity and difﬁculty level regarding DNS training principles. The participants were instructed to refrain from engaging in high-intensity anaerobic or anaerobic resistance training throughout the study period to prevent potential disruptions in the study results.

Whole body vibration group (VIBRO) WBV was performed on the Power Plate Next Generation vibration platform (Power Plate North America, Chicago, IL). All training routines were approximately 50 minutes long, commencing with 5 minutes of moderate-intensity warm-up and concluding with a cool-down period. The program consisted of 8-10 static and dynamic exercises for PS that progressively increased in difficulty and complexity. During the training process, the frequency increased from 20 to 35 Hz in the last week of the experiment; the exercise duration was from 20 - 60 seconds (in the previous week), followed by 1-minute seated rest. Moreover, the complexity and difficulty of exercise increased over the experimental period. The resting period between sets was constant from the start to the end of the training process. During the experiment, the WBV intervention group performed three weekly training sessions. The participants were advised to avoid participating in high-intensity anaerobic or anaerobic resistance training during the study to ensure that it would not interfere with the study's outcomes-no changes to trial outcomes after the trial commenced. Principles and basic procedures were adapted from previous research.

Dynamic neuromuscular stabilisation with whole body vibration group (MIX) During the two months, participants in the MIX group performed training consisting of 3 weekly sessions. The protocol consisted of a 50-minute exercise program with a 5-minute moderate-intensity warm-up and cool-down period per training session. The structural core of training included 20 minutes of WBV and 20 minutes of DNS training. Both protocols followed the previous research and training recommendations and were performed with less time and sets. Exercises with VIBRO were performed on the Power Plate Next Generation vibration platform (Power Plate North America, Chicago, IL). The program consisted of 6-8 exercises (static and dynamic) for balance and PS. Exercise progressively increases by the level of difﬁculty. During the training process, the frequency was also increased from 20 to 35 Hz in the last week of the experiment; the duration of exercise from 20 - 60 seconds (in the previous week), followed by 1-minute seated rest. The resting period between sets was constant from the start to the end of the training process. To prevent any interference with the study's results, participants were recommended to abstain from engaging in high-intensity anaerobic or anaerobic resistance training throughout the study. Basic principles and procedures were adapted from previous research. WBV is followed by 20 minutes of DNS training, including specific movement exercises according to the DNS approach accompanied by breathing, coordination, mobility, and stability core exercises and routines suggested in previous studies. During the experiment, the MIX intervention group performed three training sessions weekly.

Control group (CONTROL) The control group did not exercise or use any training intervention or other habitual training during the past two months. During this period, the control group maintained their regular daily routines without any modifications. They refrained from engaging in any form of physical activity or participating in training programs that could influence their fitness levels.

Statistical analyses G*power 3.1 power analysis software (Heinrich-Heine-University, Düsseldorf, Germany) estimated the minimum total sample size (N=140) given the critical F(3, 136)=2.67, an effect size f=0.14 (partial η2=0.02), p=0.05, 1-β=0.80, groups=4, time points=2, and correlation among the measurements=0.50. The authors presented data as means and 95% confidence intervals [95% CIs]. The Kolmogorov-Smirnov, Leven's, Box's, and Mauchly's tests confirmed the assumptions of normality, homogeneity of variances and covariances, and sphericity, respectively. General linear models (twelve separate 2x4 mixed-design analyses of covariances for each PS measure) estimated whether mean changes [95% CIs] in PS measure from initial to final testing depended on whether participants received the DNS, VIBRO, and MIX exercise program or did not (CONTROL) after controlling for mean-centered BMI. Following the time-by-group interaction effects, which revealed whether estimated changes over time depended on the participants' group (i.e., differed at least between one group-comparison pair), we computed simple effects tests to estimate mean changes over time (mean difference from initial to final testing) within the groups. The follow-up investigation proceeded with contrast analysis, which assessed the degree to which estimated mean changes of PS measures differed between the group-comparison pairs. The authors calculated the effect size for time-by-group interaction effects and simple effects using partial eta squared (partial η2: 0.01 small; 0.06 medium; 0.14 large) and Hedge's g average (Hedge'sav: <|0.20| trivial; |0.20| small; |0.50| medium; |0.80| large), respectively. The Bonferroni test corrected p-values and 95% CI; the alpha level was p≤0.05. We used SPSS version 23.0 (SPSS Inc., Chicago, IL, USA) and GraphPad Prism version 8.0 (GraphPad Software, San Diego, California, USA) to analyse and plot the data, respectively.

ELIGIBILITY:
Inclusion Criteria:

* history of neurological or musculoskeletal disorders;
* clinical conditions that could impair balance (motor disorders, medical conditions like diabetes, heart disease, stroke, issues with vision, thyroid, nerves, or blood vessels).

Exclusion Criteria:

* the absence of injuries in the past six months
* the absence of other medical conditions, including COVID-19
* no programmed physical activity in the past three months.

Ages: 21 Years to 26 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 180 (Actual)
Dates: Start 2022-02-15 (Actual); Primary Completion 2022-02-20 (Actual); Study Completion 2022-06-25 (Actual)

PRIMARY OUTCOMES:
Double-leg static postural stability sway area | 2 months
  Double leg static postural stability sway area was evaluated using a 0.5 m Footscan® plate from RSscan International, Belgium, featuring 4096 sensors and a scanning rate of up to 300 Hz. Participants completed single and double-leg tasks, each lasting 30 seconds with three trials and a two-minute break between each. During the double-leg stance, they were instructed to maintain a still, upright posture, standing comfortably with feet shoulder-width apart, barefoot, eyes open, and fixed on a cross 5 meters away at eye level on a blackboard. Arms were kept by their sides. Measurement began after a 10-second preparation period to avoid transient effects. Double-leg static postural stability sway area is analyzed in square centimeters.
Double-leg static postural stability center of force traveled way | 2 months
  Double leg static postural stability center of force traveled way was evaluated using a 0.5 m Footscan® plate from RSscan International, Belgium, featuring 4096 sensors and a scanning rate of up to 300 Hz. Participants completed single and double-leg tasks, each lasting 30 seconds with three trials and a two-minute break between each. During the double-leg stance, they were instructed to maintain a still, upright posture, standing comfortably with feet shoulder-width apart, barefoot, eyes open, and fixed on a cross 5 meters away at eye level on a blackboard. Arms were kept by their sides. Measurement began after a 10-second preparation period to avoid transient effects. Double-leg static postural stability center of force traveled way is analyzed in millimeters.
Double-leg static postural stability medio-lateral displacement | 2 months
  Double leg static postural stability medio-lateral displacement was evaluated using a 0.5 m Footscan® plate from RSscan International, Belgium, featuring 4096 sensors and a scanning rate of up to 300 Hz. Participants completed single and double-leg tasks, each lasting 30 seconds with three trials and a two-minute break between each. During the double-leg stance, they were instructed to maintain a still, upright posture, standing comfortably with feet shoulder-width apart, barefoot, eyes open, and fixed on a cross 5 meters away at eye level on a blackboard. Arms were kept by their sides. Measurement began after a 10-second preparation period to avoid transient effects. Double-leg static postural stability medio-lateral displacement is analyzed in millimeters.
Double-leg static postural stability anterior-posterior displacement | 2 months
  Double leg static postural stability anterior-posterior displacement was evaluated using a 0.5 m Footscan® plate from RSscan International, Belgium, featuring 4096 sensors and a scanning rate of up to 300 Hz. Participants completed single and double-leg tasks, each lasting 30 seconds with three trials and a two-minute break between each. During the double-leg stance, they were instructed to maintain a still, upright posture, standing comfortably with feet shoulder-width apart, barefoot, eyes open, and fixed on a cross 5 meters away at eye level on a blackboard. Arms were kept by their sides. Measurement began after a 10-second preparation period to avoid transient effects. Double-leg static postural stability anterior-posterior displacement is analyzed in millimeters.
Single-leg static postural stability sway area | 2 months
  Single leg static postural stability sway area was evaluated using a 0.5 m Footscan® plate from RSscan International, Belgium, equipped with 4096 sensors and a scanning rate of up to 300 Hz. During the single-limb stance test, participants balanced on one foot, aligning it forward with reference lines in the frontal and sagittal planes. The swinging leg was flexed at the hip and knee to about 90 degrees, while arms hung naturally at their sides. Participants were instructed to maintain a steady posture, focusing on a point 65 centimeters away on the wall. The order of testing between legs was randomized. Measurement began after a 5-second preparation period. Single-leg static postural stability sway area is analyzed in square centimeters..
Single-leg static postural stability center of force traveled way | 2 months
  Single leg static postural stability center of force traveled way was evaluated using a 0.5 m Footscan® plate from RSscan International, Belgium, equipped with 4096 sensors and a scanning rate of up to 300 Hz. During the single-limb stance test, participants balanced on one foot, aligning it forward with reference lines in the frontal and sagittal planes. The swinging leg was flexed at the hip and knee to about 90 degrees, while arms hung naturally at their sides. Participants were instructed to maintain a steady posture, focusing on a point 65 centimeters away on the wall. The order of testing between legs was randomized. Measurement began after a 5-second preparation period. Single-leg static postural stability center of force traveled way is analyzed in millimeters.
Single-leg static postural stability anterior-posterior displacement | 2 months
  Single leg static postural stability anterior-posterior displacement was evaluated using a 0.5 m Footscan® plate from RSscan International, Belgium, equipped with 4096 sensors and a scanning rate of up to 300 Hz. During the single-limb stance test, participants balanced on one foot, aligning it forward with reference lines in the frontal and sagittal planes. The swinging leg was flexed at the hip and knee to about 90 degrees, while arms hung naturally at their sides. Participants were instructed to maintain a steady posture, focusing on a point 65 centimeters away on the wall. The order of testing between legs was randomized. Measurement began after a 5-second preparation period. Single-leg static postural stability anterior-posterior displacement is analyzed in millimeters.
Single-leg static postural stability medio-lateral displacement | 2 months
  Single leg static postural stability medio-lateral displacement was evaluated using a 0.5 m Footscan® plate from RSscan International, Belgium, equipped with 4096 sensors and a scanning rate of up to 300 Hz. During the single-limb stance test, participants balanced on one foot, aligning it forward with reference lines in the frontal and sagittal planes. The swinging leg was flexed at the hip and knee to about 90 degrees, while arms hung naturally at their sides. Participants were instructed to maintain a steady posture, focusing on a point 65 centimeters away on the wall. The order of testing between legs was randomized. Measurement began after a 5-second preparation period. Single-leg static postural stability medio-lateral displacement is analyzed in millimeters.

SECONDARY OUTCOMES:
Sex | 2 months
  The sex of the participants is recorded at the start of the study.
Date of birth | 2 months
  The participant's date of birth is collected in order to calculate his age in years.
Weight | 2 months
  The weight of the participants is analyzed in kilograms.
Height | 2 months
  The height of the subject is determined in meters.
Body Mass Index (BMI) | 2 months
  The participant's BMI is calculated from his height and weight.
Adherence | 2 months
  Adherence to the program is calculated from the record of the percentage of attendance at the intervention sessions.

CONTACTS AND LOCATIONS:
Overall Officials: Dragan Marinkovic, MSc, Principal Investigator — University of Novi Sad, Faculty of Sport and Physical Education
Locations (1):
- Faculty of sport and Physical Education, University of Novi Sad, Novi Sad, Vojvodina, Serbia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Marinkovic D, Macak D, Madic DM, Sporis G, Kuvacic D, Jasic D, Petric V, Spehnjak M, Projovic A, Gojkovic Z. Effect of Neuromuscular Training Program on Quality of Life After COVID-19 Lockdown Among Young Healthy Participants: A Randomized Controlled Trial. Front Psychol. 2022 Apr 12;13:844678. doi: 10.3389/fpsyg.2022.844678. eCollection 2022. PMID 35496239

DOCUMENTS (2):
  • Study Protocol (2024-02-19): https://cdn.clinicaltrials.gov/large-docs/02/NCT06294002/Prot_000.pdf
  • Informed Consent Form (2024-02-19): https://cdn.clinicaltrials.gov/large-docs/02/NCT06294002/ICF_001.pdf